CLINICAL TRIAL: NCT06862141
Title: Bendable Suction Ureteral Access Sheath Versus Conventional Ureteral Access Sheath in Treatment of Renal Stones Using Flexible Ureteroscopy: a Randomized Clinical Trial
Brief Title: Bendable Suction Ureteral Access Sheath Versus Conventional Ureteral Access Sheath in Management of Renal Stones Using Flexible Ureteroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Abdelazez Anwar Nuser, Teaching assistant of urology , urology department , menoufia university, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FANS protocol
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Nephrolithiasis; Flexible Ureteroscopy
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- bendable suction ureteral access sheath (Experimental): this group will undergo flexible ureteroscopy using bendable suction ureteral access sheath
  Interventions: Device: bendable suction ureteral access sheath
- conventional ureteral access sheath (Experimental): this group will undergo flexible ureteroscopy using conventional ureteral access sheath
  Interventions: Device: conventional suction ureteral access sheath

INTERVENTIONS:
Device: bendable suction ureteral access sheath — flexible ureteroscopy will be done using bendable suction ureteral access sheath
  Arms: bendable suction ureteral access sheath
Device: conventional suction ureteral access sheath — flexible ureteroscopy will be done using conventional suction ureteral access sheath
  Arms: conventional ureteral access sheath

SUMMARY:
Urinary calculus is a globally recognized urological condition, with prevalence rates ranging from 1% to 13% across different geographical regions (1) Therapeutic approaches for renal calculi encompass extracorporeal shock wave lithotripsy (ESWL) and minimally invasive endoscopic surgical techniques, such as percutaneous nephrolithotomy (PCNL) and retrograde intrarenal surgery (RIRS). Treatment plans depend on the characteristics of calculi, patient factors, surgeon experience and the condition of medical centers. According to the guidelines of American Urologic Association (AUA) and European Association of Urology (EAU), patients with a burden of less than 20 mm in kidney calculi can choose RIRS as the frst-line surgical treatment with good stone-free rate (SFR). (2, 3) The application of RIRS for urinary stones has increased signifcantly, and the indications have expanded due to developments in minimally invasive technology and equipment. (4) With the development of stone retrieval devices and miniaturized fexible ureteroscopes, RIRS is more widely used for treating renal calculi, even for high burden stones. (5, 6) The application of ureteral access sheath (UAS) in RIRS can improve surgical vision, reduce intrarenal pressure (IRP), and decrease postoperative infectious complications. (7-9) Several reports have demonstrated the superiority of suctioning UAS, including shorter operation time, higher SFR and lower incidence of infectious complications compared with traditional ureteral access sheath, but none of these suctioning UAS can reach the renal calyces. (10-12)

A novel tip-flexible suctioning ureteral access sheath with flexible terminal was designed, which delivered the tip of the ureteral access sheath to renal calyces. However, data comparing novel tip-flexible suctioning ureteral access and traditional ureteral access sheath is lacking in RIRS.

Therefore, we designed a prospective controlled analysis to compare the efficacy and safety of novel tip-flexible suctioning ureteral access sheath and traditional ureteral access sheath combined with flexible ureteroscope (FURS) in treating renal calculi.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Radiologically confirmed renal stones (e.g., CT, ultrasound, or X-ray).
* Stone size within a specific range (e.g., 5-20 mm).
* Indication for Treatment: patients indicated for flexible ureteroscopy due to renal stones.
* Anatomical Suitability: normal or mildly altered renal anatomy that allows safe use of the access sheath.
* Willingness to participate and provide written informed consent.

Exclusion Criteria:

* - Medical Conditions: Active urinary tract infection (UTI) or sepsis. Coagulopathy or inability to discontinue anticoagulation therapy. Significant comorbidities (e.g., severe cardiopulmonary disease). Pregnancy: Pregnant or breastfeeding individuals.
* Anatomical or Surgical Factors:

Severe ureteral stricture or obstruction preventing sheath placement. Congenital abnormalities affecting the urinary tract. - Stone Factors: Stones larger than the sheath's operational limit (e.g., >20 mm). Multiple stones in different calyces that cannot be accessed in one session.

- Previous Treatment: Recent (<6 weeks) or repeated interventions for the same stones (e.g., prior lithotripsy or ureteroscopy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Immediate stone free rate | one day postoperative
  measured by the number of cases has the status of No residual stone or stone fragments less than 2 mm on low-dose CT scan at postoperative day 1 are defined as stone free.

SECONDARY OUTCOMES:
3 month stone free rate | 3 months postoperatively
  measured by number of cases has the status of No residual stone or stone fragments less than 2 mm on low-dose CT scan at postoperative day 1 are defined as stone free.
duration of hospital stay | 2 weeks
  measured by number of days from the day of operation till the discharge day
secondary intervention | 3 months
  measured by the number of interventions received post randomization
complications | 3 months
  measured by the number of complications experienced by the patients
costs | 3 months postoperatively
  measured by the total costs of patient during hospitalization and up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Menoufia University, Shebin Elkom, Menoufia, Egypt